CLINICAL TRIAL: NCT05722743
Title: Improving Person-Environment Fit of Community-Residing Older Adults With Dementia
Brief Title: Person-Environment Fit for Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth K Rhodus (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Elizabeth K Rhodus, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 72893; 1K23AG075262-01A1 (NIH)
Record Dates: First submitted 2022-12-27; First posted 2023-02-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Dementia Alzheimers; Alzheimer Disease
Keywords: Behavioral; Occupational therapy; Alzheimer's disease and related dementias; Telehealth; Caregiver
MeSH Terms: conditions — Alzheimer Disease; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Harmony at HOME (Experimental): Participants in this group will receive the Harmony at HOME intervention.
  Interventions: Behavioral: Harmony at HOME
- National Institute on Aging Program (Active Comparator): Participants in this group will receive the National Institute on Aging education.
  Interventions: Behavioral: National Institute on Aging Program

INTERVENTIONS:
Behavioral: Harmony at HOME — The Harmony at HOME (Help Online Modifying the Environment) intervention builds on prior successful foundations of dementia care interventions with a novel approach combining remote implementation, antecedent education, and home environment intervention. The intervention will teach caregivers how to 1) assess the home environment as an antecedent to behavior for the person with ADRD, and 2) design and implement individualized environmental modification through an environmental cueing approach to address the needs of the person with ADRD in a supportive environment.
  Arms: Harmony at HOME
Behavioral: National Institute on Aging Program — Standard of care will address behaviors and psychiatric symptoms of dementia (BPSD) for persons with ADRD, as recommended by their medical provider. Caregivers will receive training regarding home safety via a home safety handout based on National Institutes on Aging "Home Safety and Alzheimer's Disease" webpage.
  Arms: National Institute on Aging Program

SUMMARY:
This trial will assess feasibility of a non-pharmacological intervention for persons living with Alzheimer's disease and related dementias (ADRD) to improve behavioral and psychiatric symptoms of dementia and functional performance.

Using a two-arm, prospective randomized controlled trial, 38 dyads (person with ADRD and caregiver) will complete an 8-week telehealth occupational therapy intervention provided via Zoom with caregivers and persons with dementia or receive an active control with 8 telehealth sessions to discuss publicly available caregiver education with a non-clinical research assistant.

ELIGIBILITY:
Inclusion Criteria: Participants with Dementia

* Men or women aged 60-99, inclusive.
* Living at home in the community with one primary caregiver.
* Diagnosis or probably diagnosis of dementia (confirmed by Clinical Dementia Rating Scale score of 1.0+)
* If on psychotropic medication, they are at a point where dosage and treatment are stabilized for the duration of the study.
* Functional sensory abilities with or without aids (hearing, vision, smell, touch, taste)
* Caregiver report of challenges related to behaviors within 4 weeks of study enrollment.
* Caregiver willing to participate throughout duration of study.
* Contact with University of Kentucky Alzheimer's Disease Research Center or Kentucky Neuroscience Institute medical provider within 12 months of study recruitment.

Inclusion Criteria: Caregiver for Participants with Dementia

* Men or women aged 21-99, inclusive.
* Willingness to participate in study and implement recommended data collection tools.
* English speaking, able to read and write.
* Ability to retrieve and send mail.

Exclusion Criteria: Participants with Dementia

* Unstable medical conditions within one month prior to screening visit such as poorly controlled blood pressure, diabetes, current cancer diagnosis, or breathing problems, etc.
* Wheelchair or bed bound.
* Residence in skilled nursing facility or facility-based care.
* Caregiver report of physically violent behaviors.
* Initiation of antipsychotic medication within 4 weeks prior to screening or unpredictable use of such medications
* Diagnosis of profound or total sensory altering disorders including macular degeneration, legal blindness, total deafness, severe peripheral neuropathy, anosmia.
* Major depression in past 12 months (DSM-IV criteria), major mental illness such as schizophrenia, bipolar disorder, personality disorders, or recent (in past 12 months) alcohol or substance abuse.
* Major infection within 4 weeks prior to the Baseline Visit.

Exclusion Criteria: Caregiver for Participant with Dementia:

• Diagnosis of mild cognitive impairment or dementia.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Change in patient performance as measured by Canadian Occupational Performance Measure (COPM) | 13weeks (baseline, post-intervention, follow up)
  Criterion-referenced interview of patient performance with caregiver The COPM is a reliable and validated measure of performance in primary daily activities (self-care, leisure, productivity) with dyad-caregiver rated of performance and satisfaction. Scores are determined on a likert scale of 1-10 with 1 being lowest and 10 indicating highest of the topic of the question.
Caregiver satisfaction of patient performance [Feasibility] | 13 weeks (baseline, post intervention, follow up)
  The primary outcome analysis is the feasibility of implementation as measured by caregiver satisfaction. The Canadian Occupational Performance Measure will measure caregiver satisfaction of patient performance, high scores indicate higher levels of satisfaction. Range 0-10.

SECONDARY OUTCOMES:
Zarit Caregiver Burden Scale | 13 weeks (baseline, post intervention, follow up)
  22-item survey, caregiver rates self-perceived level of burden on 5-point Likert scale. The social context of the person with ADRD will be described through analysis of caregiver demographics and rate of caregiver burden measured. Higher scores indicate greater burden. Range of 0-88 points. A score of 17 or more was considered high burden.
Neuropsychiatric Inventory Questionnaire (NPI-Q) | 13 weeks (baseline, post intervention, follow up)
  The NPI-Q is commonly used as an assessment of behavioral and psychiatric symptoms of dementia in older adults diagnosed with mild cognitive impairment or dementia, internationally, with high reliability and validity. Assessment includes 12 behavioral and psychiatric domains which are rated by caregiver as present or absent (yes/no). Caregivers further rate severity of present behavioral domains. The severity score is summed to yield a total as a measure of BPSD burden. Higher scores indicate higher levels of behavior symptom severity and/or distress. Range 0-36
Functional Behavior Profile (FBP) | 13 weeks (baseline, post intervention, follow up)
  Criterion-referenced survey completed by caregiver. The FBP has been established as a reliable and valid measure of task performance, social interaction, and problem solving with adults with ADRD. Item responses range from 0 to 4, with higher scores indicating better performance (maximum score 108).

OTHER OUTCOMES:
Home Occupational Environment Assessment (HOEA) | 1 time (baseline)
  35-item survey completed by caregiver regarding home environment. Allows the caregiver to systematically assess the home environment including accessibility, sanitation, food storage, safety, and sensorial stimulation. Scores range 0-105 with higher scores indicating worse outcomes.
Adult Sensory Profile (ASP) | 1 time (baseline)
  Norm-referenced, 60-item survey completed by caregiver. The caregiver will complete the Adult Sensory Profile as proxy for person with ADRD. This is a valid and reliable 60-question assessment to determine sensory simulation preference and neurological ability for processing sensory simulation. This assessment is not based on a range of scores but normative values. Results can be more than or less than normative values.
Clinical Dementia Rating Scale (CDR-SUM) | 1 time (baseline)
  The Clinical Dementia Rating (CDR) sum of boxes, a valid and reliable measure, will determine severity of cognitive impairment. Six cognitive domains are assessed in CDR (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care) with feedback from patient performance and caregiver result, and results are scored by a trained professional. Range 0-18, higher scores indicate higher levels of cognitive impairment.
Digital Biomarker of psychophysiological response to environment: heart rate variability | Device worn by patient for 7 consecutive days
  Empatica wearable wrist device Assessment of stress-related biomarkers will measure heart rate variability in beats per minute.
Digital Biomarker of psychophysiological response to environment: electrodermal activity | Device worn by patient for 7 consecutive days
  Empatica wearable wrist device Assessment of stress-related biomarkers will measure electrical conductance at the surface of the skin. Skin conductance is measured in units of microsiemens, with normal human EDA ranging from 1 to 20 microsiemens.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rhodus, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT05722743/ICF_000.pdf